CLINICAL TRIAL: NCT00593827
Title: Phase II Randomized Trial of Weekly and Every 3-week Ixabepilone in Metastatic Breast Cancer (MBC) Patients
Brief Title: Phase II Trial of Weekly or Every 3-week Ixabepilone for Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: US Oncology Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-132; USOR 06-106
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Results first posted 2012-05-25 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): ixabepilone 16 mg/m^2 weekly for 3 weeks followed by 1 week rest
  Interventions: Drug: Ixabepilone
- Arm 2 (Active Comparator): ixabepilone 40 mg/m^2 every 3 weeks
  Interventions: Drug: Ixabepilone

INTERVENTIONS:
Drug: Ixabepilone — Injection, IV, Until progressive disease or intolerable toxicity Ixabepilone 16 mg/m^2 was administered as a 1-hour IV continuous infusion on Days 1, 8, and 15 in a 28-day cycle until progressive disease or intolerable toxicity.
  Other Names: IXEMPRA; BMS-247550
  Arms: Arm 1
Drug: Ixabepilone — Injection, IV, Until progressive disease or intolerable toxicity Ixabepilone 40 mg/m^2 was administered as a 3-hour IV infusion on Day 1 of each 21-day cycle provided the subject met the retreatment criteria.
  Other Names: IXEMPRA; BMS-247550
  Arms: Arm 2

SUMMARY:
The purpose of this study was to determine the effects of the weekly regimen of ixabepilone dosing compared to the once every 3 week dosing regimen in participants with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has MBC that is measurable by RECIST or has nonmeasurable disease with serum CA27.29 (or CA15.3) ≥ 50
* Has Human Epidermal Growth Factor Receptor 2 (HER2) negative breast cancer
* Prior chemotherapy is permitted with no limit on the number of prior regimens
* Two weeks or more have elapsed since last chemotherapy or radiation treatment
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-2
* Is female, ≥ 18 yrs of age
* Protocol defined appropriate laboratory values
* Negative pregnancy test within 7 calendar days prior to registration
* Has signed a patient informed consent

Exclusion Criteria:

* Had prior treatment with ixabepilone or other epothilones
* Has HER2+ disease
* Has a known, prior, severe (National Cancer Institute Common Terminology Criteria Adverse Events [NCI CTCAE] Grade 3-4) history of hypersensitivity reaction to a drug formulated in Cremophor ® EL (polyoxyethylated castor oil)
* Is receiving concurrent immunotherapy, hormonal therapy or radiation therapy
* Is receiving concurrent investigational therapy or has received such therapy within the past 30 days
* Has peripheral neuropathy > Grade 1
* Has evidence of central nervous system (CNS) involvement requiring radiation or steroid treatment. Participants with stable brain metastases who are off steroids at least 2 weeks are eligible
* Is pregnant or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2008-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (57):
- United States (57):
  - Birmingham Hematology & Oncology Associates Llc, Birmingham, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Northern Arizona Hematology & Oncology Associates, Sedona, Arizona
  - Arizona Oncology Associates D.B.A. Hematology Oncology, Tucson, Arizona
  - Southwest Cancer Care, Murrieta, California
  - Florida Cancer Institute, Hudson, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers Of Florida, P.A, Ocoee, Florida
  - Cancer Care & Hematology Specialists Of Chicagoland, Niles, Illinois
  - Central Indiana Cancer Centers, Carmel, Indiana
  - Hope Center, Terre Haute, Indiana
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Alliance Hematology Oncology, Pa, Westminster, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Kansas City Cancer Center, Llc, Kansas City, Missouri
  - Arch Medical Services, Inc., St Louis, Missouri
  - Comprehensive Cancer Center Of Nevada, Henderson, Nevada
  - Hematology-Oncology Assoc. Of Northern Nj, Pa, Morristown, New Jersey
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, P.C., Amsterdam, New York
  - Interlakes Oncology & Hematology, P.C., Rochester, New York
  - Regional Cancer Care, Durham, North Carolina
  - Raleigh Hematology Oncology Associates, Raleigh, North Carolina
  - Cancer Centers Of The Carolinas, Greenville, South Carolina
  - Texas Cancer Center, Arlington, Texas
  - Texas Oncology-Central Austin Cancer Center, Austin, Texas
  - Mamie Mcfaddin Ward Cancer Center Texas Oncology, Beaumont, Texas
  - Texas Oncology, Bedord, Texas
  - Texas Cancer Center At Medical City, Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology/Methodist Charlton Cancer Ctr, Dallas, Texas
  - Baylor Sammons Cancer Ctr, Dallas, Texas
  - Texas Oncology Sammons Cancer Center, Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - Texas Oncology, Fort Worth, Texas
  - Texas Oncology, Garland, Texas
  - Texas Oncology, Houston, Texas
  - Texas Oncology - Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cancer Center, Longview, Texas
  - South Texas Cancer Center, McAllen, Texas
  - Texas Cancer Center Of Mesquite, Mesquite, Texas
  - Texas Oncology, Pa, Midland, Texas
  - Texas Oncology - Odessa, Odessa, Texas
  - Paris Regional Cancer Center Lab, Paris, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology Cancer Center - Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer Care And Research Center, Waco, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - Oncology & Hematology Associates Of Southwest Virginia, Inc., Salem, Virginia
  - Puget Sound Cancer Centers, Edmonds, Washington
  - Puget Sound Cancer Centers, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Evergreen Hematology And Oncology, Spokane, Washington
  - Northwest Cancer Specialists, Pc, Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 176 participants were enrolled by 55 sites in the United States over a period of 12 months.
Pre-assignment Details: All the 176 enrolled participants were randomized. Of the 5 participants who did not receive treatment, 2 were due to disease progression, 1 on participant request, and 2 due to other reasons.
Groups:
- Ixabepilone 16 mg/m^2: ixabepilone 16 mg/m^2 weekly for 3 weeks followed by 1 week rest
- Ixabepilone 40 mg/m^2: ixabepilone 40 mg/m^2 every 3 weeks
Period: Overall Study
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2
Started | 85 (Intent-to-Treat (ITT) Population: Participants who were randomized (eligible and ineligible).) | 91 (ITT Population: Participants who were randomized (eligible and ineligible).)
Safety Population | 82 (Participants (eligible and ineligible) who received at least 1 dose of study drug.) | 89 (Participants (eligible and ineligible) who received at least 1 dose of study drug.)
Evaluable Population | 79 (Treated participants with CR, PR, SD, PD, or NE response. Refer outcome measure 3 and 4 for details.) | 89 (Treated participants with CR, PR, SD, PD, or NE response. Refer outcome measure 3 and 4 for details.)
Completed | 85 (Completed=off-study (Major reasons: Adverse events (AE)=15; disease progression=76; not treated=3).) | 89 (Completed=off-study (Major reasons: AEs=30; disease progression=55; not treated=2).)
Not Completed | 0 | 2
Not completed — On Active Treatment/Pending | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2 | Total
Number analyzed (Participants) | 85 | 91 | 176
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (11.4) | 58.7 (10.4) | 59.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 91 | 176
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 69 | 70 | 139
  African American | 9 | 10 | 19
  Hispanic | 6 | 11 | 17
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: Participants]
  United States | 85 | 91 | 176
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: Participants] — The ECOG PS is used to assess disease severity. A score of 0 is normal activity; 1 is symptoms, but fully ambulatory; 2 is symptomatic, but in bed < 50% of the day; 3 is needs to be in bed > 50% of the day, but not bedridden; 4 is unable to get out of bed; 5 is dead.
  Participants
    0=normal activity | 39 | 43 | 82
    1=symptoms, but fully ambulatory | 40 | 43 | 83
    2=symptomatic, but in bed < 50% of the day | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) at 6 Months (6-month PFS Rate): Proportion of Participants Progression Free at 6 Months
Description: PFS at 6 months was defined as proportion of participants who neither progressed nor died before 6 months. Computed using Kaplan-Meier estimates.
Time Frame: From the date of randomization to 6-months on study
Population: ITT population: Participants who were randomized on the study (eligible and ineligible).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 85 | 91
Percentage of Participants | 28.6 [18.9 to 38.9] | 42.7 [31.5 to 53.5]
Statistical Analysis 1: Comparison: Ixabepilone 16 mg/m^2 vs Ixabepilone 40 mg/m^2; Test type: Superiority or Other; p = 0.03, Log Rank

2. Secondary Outcome: Median Progression Free Survival
Description: PFS is defined as time interval from the date of randomization to the date of (first) progression or date of death. Participants who progressed or died were counted as events. Participants lost to follow-up were censored as of the last date of contact. Participants who started a new treatment before they progressed were censored as of the date of start of the new treatment. Participants who had not progressed or died were censored at the date of last follow-up. PFS (months) = (End date - date of randomization + 1)/30.4375.
Time Frame: From the date of randomization to date of progression, death, or last tumor assessment (maximum participant PFS of 25.7 months)
Population: ITT population: Participants who were randomized on the study (eligible and ineligible).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 85 | 91
Months | 2.9 [2.7 to 5.1] | 5.3 [3.8 to 6.2]
Statistical Analysis 1: Comparison: Ixabepilone 16 mg/m^2 vs Ixabepilone 40 mg/m^2; Test type: Superiority or Other; p = 0.05, Log Rank

3. Secondary Outcome: Overall Response Rate (ORR) Based on Response Criteria in Solid Tumors [RECIST]
Description: ORR is defined as the proportion of responders (complete response [CR] + partial response [PR] in participants with measurable disease) in that arm among all randomized participants.
  CR: Disappearance of all evidence of target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (LD) of all target lesions.
  Measurable disease: Lesions that can be accurately measured in at least one dimension (LD to be recorded) as ≥20 mm with conventional techniques (computed tomography [CT], magnetic resonance imaging [MRI], X-ray) or as ≥10 mm with spiral CT scan.
Time Frame: Assessed at 12-week intervals until disease progression (to a maximum follow-up for tumor response of 26.3 months)
Population: Evaluable population-All treated participants with CR, PR, stable disease (SD), progressive disease (PD), or nonevaluable (NE) response and who had received at least 1 dose of study drug. Please refer outcome measure 4 for explanation of SD, PD, and NE.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 79 | 89
Percentage of Participants | 7.6 [2.8 to 15.8] | 13.5 [7.2 to 22.4]

4. Secondary Outcome: Best Response as Assessed With RECIST
Description: Determined based on the sequence of disease status with corresponding best response. PD=At least a 20% increase in the sum of LD of target lesions in reference to the smallest sum LD recorded or the appearance of 1 or more new lesions; SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD in reference to the smallest sum LD. NE=Participants who discontinued treatment secondary to toxicity or died (either before completion of 1 treatment cycle). Please refer outcome measure 3 for explanation of CR and PR. CR+PR+SD=overall disease control.
Time Frame: Assessed at 12-week intervals until disease progression (to a maximum follow-up for tumor response of 26.3 months)
Population: Evaluable population: All treated participants with CR, PR, SD, PD, or NE response and who had received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 79 | 89
Percentage of Participants
  CR | 0 [NA to NA] — No participants had CR. | 1.1 [0.0 to 6.1]
  PR | 7.6 [2.8 to 15.8] | 12.4 [6.3 to 21.0]
  SD | 40.5 [29.6 to 52.1] | 44.9 [34.4 to 55.9]
  SD>=6 months | 19.0 [11.0 to 29.4] | 15.7 [8.9 to 25.0]
  PD | 41.8 [30.8 to 53.4] | 29.2 [20.1 to 39.8]
  NE | 10.1 [4.5 to 19.0] | 12.4 [6.3 to 21.0]
  CR+PR+SD>=6 mos | 26.6 [17.3 to 37.7] | 29.2 [20.1 to 39.8]

5. Secondary Outcome: Overall Survival (OS)
Description: Survival was measured as the date of randomization to the date of death. Participants who were alive at the time of the database lock or lost to follow-up were censored at the last known alive date. The distribution of overall survival was analyzed via the Kaplan Meier method in each arm.
  Survival time (months) = (End date - date of randomization + 1)/30.4375
Time Frame: From the date of randomization to date of death (maximum participant OS of 26.3 months)
Population: ITT population: Participants who were randomized on the study (eligible and ineligible).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 85 | 91
Months | 13.9 [12.1 to 15.7] | 16.1 [10.3 to NA] — Insufficient number of participants with an event were available to estimate the upper limit of the confidence interval.
Statistical Analysis 1: Comparison: Ixabepilone 16 mg/m^2 vs Ixabepilone 40 mg/m^2; Test type: Superiority or Other; p = 0.11, Log Rank

6. Secondary Outcome: Time to Response
Description: Time to response is defined as the time from the start of treatment until the first (confirmed) CR or PR was recorded. Time to response was computed only for participants whose best response was PR or CR.
  CR: Disappearance of all target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (LD) of all target lesions with reference to the baseline sum LD.
Time Frame: From the date of first dose to date of first PR or CR assessment ( maximum participant time to response of 8.3 months)
Population: ITT population with CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 6 | 12
Months | 2.5 [1.7 to 8.3] | 2.8 [2.0 to 8.1]

7. Secondary Outcome: Duration of Response
Description: Duration of overall response was defined as the period from the time first PR or CR was recorded until the first date of documented PD or death. Duration of response was computed for participants whose best response was either PR or CR. Participants who neither relapsed nor died were censored on the date of their last tumor assessment. Kaplan-Meier method was used to estimate the duration of response. Refer to outcome measures 3 and 4 for CR, PR, and PD.
Time Frame: From the date of first PR or CR assessment to date of progression, death, or last tumor assessment (maximum participant duration of response of 17.4 months)
Population: ITT population with CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 6 | 12
Months | 6.2 [3.3 to NA] — Insufficient number of participants with an event were available to estimate the upper limit of the confidence interval. | 6.3 [4.1 to 17.3]

8. Other Pre Specified Outcome: Number of Participants With Death as Outcome, Treatment-related (TR) Deaths, SAEs, TR SAEs, Adverse Events (AEs) Leading to Discontinuation, AEs, TR AEs, GR 3-4 AEs, TR GR 3-4 AEs, Drug-related (DR) Peripheral Neuropathy, Neutropenia, Alopecia
Description: An AE is any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical event that at any dose: results in death, persistent or significant disability/incapacity, drug dependency or abuse; is life-threatening, an important medical event, a congenital anomaly/birth defect; requires inpatient hospitalization; or prolongs existing hospitalization. Treatment related=possibly, probably, or certainly related to and of unknown relationship to study treatment. GR=Grade.
Time Frame: Assessed from the date of first dose until at least 30 days after the last dose of study drug. Median time on study therapy was 12 weeks (range: 4-60 weeks for 16 mg/m^2 arm; 3-87 weeks for 40 mg/m^2 arm).
Population: ITT population: Participants randomized on the study (eligible and ineligible). AEs, AEs leading to death and GR 3-4 AEs: Safety population-Participants who received atleast 1 dose of study drug).
  AEs leading to death: For 4 participants in Arm 1 and both participants in Arm 2, the reported AE term was "disease progression."
Measure: Number; unit: Participants
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 85 | 91
Participants
  Deaths (All) | 55 | 48
  Treatment-related deaths | 0 | 0
  AEs leading to death (n=82; n=89) | 7 | 2
  At least 1 SAE | 25 | 30
  At least 1 study-related SAE | 5 | 17
  AEs leading to discontinuation | 15 | 30
  At least 1 AE (n=82; n=89) | 82 | 89
  At least 1 study-related AEs | 69 | 84
  At least 1 GR 3 and 4 AEs (n=82; n=89) | 34 | 69
  At least 1 study-related GR 3 and 4 AEs | 23 | 61
  Drug-related peripheral neuropathy (All) | 26 | 38
  GR 1 and 2 drug-related peripheral neuropathy | 19 | 24
  GR 3 drug-related peripheral neuropathy | 6 | 14
  GR 4 drug-related peripheral neuropathy | 1 | 0
  Drug-related neutropenia (All) | 15 | 47
  GR 1 and 2 drug-related neutropenia | 10 | 13
  GR 3 drug-related neutropenia | 3 | 18
  GR 4 drug-related neutropenia | 2 | 16
  Drug-related alopecia (All) | 21 | 54
  GR 1 and 2 drug-related alopecia | 21 | 54

9. Secondary Outcome: Incidence of All Grades of Peripheral Neuropathy
Description: All events of peripheral neuropathy were assessed and graded per National Cancer Institute (NCI) Common Terminology Criteria Adverse Events (CTCAE)Version 3. CTC Grade (GR) 1=Mild; GR2=Moderate; GR3=Severe or medically significant, not immediately life-threatening; and GR4=Life-threatening. All treatment-related and not related Neuropathy and Peripheral Neuropathy were included; serious adverse events (SAEs) were not included.
Time Frame: Assessed from the date of first study dose until at least 30 days after the last dose of study drug. Median time on study therapy was 12 weeks (range: 4-60 weeks for 16 mg/m^2 arm; 3-87 weeks for 40 mg/m^2 arm).
Population: Safety population.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 82 | 89
Participants
  All | 26 | 39
  Grade 1 | 9 | 15
  Grade 2 | 10 | 10
  Grade 3 | 6 | 14
  Grade 4 | 1 | 0

ADVERSE EVENTS:
Time Frame: From the date of first study dose until at least 30 days after the last dose of study drug. Median time on study therapy was 12 weeks (range: 4-60 weeks for 16 mg/m2 arm; 3-87 weeks for 40 mg/m2 arm).
Description: AEs and other symptoms were graded according to the CTCAE Version 3.0 and categorized according to Medical Dictionary for Regulatory Activities (MedDRA) Version 14.1.
Arm/Group | Ixabepilone 16 mg/m^2 | Ixabepilone 40 mg/m^2
Serious Adverse Events (participants affected / at risk) | 25/82 | 30/89
Other Adverse Events (participants affected / at risk) | 82/82 | 89/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone 16 mg/m^2 (N=82) | Ixabepilone 40 mg/m^2 (N=89)
neutropenia (Blood and lymphatic system disorders) | 1 | 5
anemia (Blood and lymphatic system disorders) | 1 | 1
thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
tachycardia (Cardiac disorders) | 3 | 1
fibrillation atrial (Cardiac disorders) | 0 | 1
supraventricular tachycardia (Cardiac disorders) | 1 | 0
ventricular tachycardia (Cardiac disorders) | 1 | 0
angina attack (Cardiac disorders) | 0 | 1
congestive heart failure (Cardiac disorders) | 0 | 1
flutter atrial (Cardiac disorders) | 0 | 1
myocardial infarction (Cardiac disorders) | 0 | 1
arrest cardiac (Cardiac disorders) | 1 | 0
cardiopulmonary arrest (Cardiac disorders) | 1 | 0
hypotension (Vascular disorders) | 1 | 0
weakness (General disorders) | 1 | 2
dehydration (Metabolism and nutrition disorders) | 2 | 9
vomiting (Gastrointestinal disorders) | 3 | 6
nausea (Gastrointestinal disorders) | 1 | 2
diarrhea (Gastrointestinal disorders) | 0 | 2
gastroparesis (Gastrointestinal disorders) | 0 | 1
ileus (Gastrointestinal disorders) | 0 | 1
mucositis (Gastrointestinal disorders) | 0 | 1
abdominal pain (Gastrointestinal disorders) | 1 | 0
colitis (Gastrointestinal disorders) | 1 | 0
anorexia (Metabolism and nutrition disorders) | 1 | 0
diverticulitis (Infections and infestations) | 1 | 0
electrolyte abnormality (Metabolism and nutrition disorders) | 1 | 0
gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0
hematoma (Vascular disorders) | 1 | 0
febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
infection bacterial (Infections and infestations) | 1 | 4
sepsis (Infections and infestations) | 0 | 1
abscess (Infections and infestations) | 2 | 0
meningitis (Infections and infestations) | 1 | 0
fever (General disorders) | 0 | 2
edema (General disorders) | 1 | 1
hypokalemia (Metabolism and nutrition disorders) | 0 | 1
glucose blood increased (Investigations) | 0 | 1
hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 3
fracture (Injury, poisoning and procedural complications) | 0 | 2
fracture pathological (Musculoskeletal and connective tissue disorders) | 0 | 1
pain bone (Musculoskeletal and connective tissue disorders) | 0 | 1
neuropathy peripheral (Nervous system disorders) | 0 | 2
lethargy (Nervous system disorders) | 0 | 1
dizziness (Nervous system disorders) | 1 | 0
neuropathy (Nervous system disorders) | 1 | 0
pain (General disorders) | 1 | 2
chest pain (General disorders) | 0 | 2
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 6 | 1
effusion pleural (Respiratory, thoracic and mediastinal disorders) | 1 | 1
pneumonia (Infections and infestations) | 1 | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
distress respiratory (Respiratory, thoracic and mediastinal disorders) | 2 | 0
embolus pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 0
failure respiratory (Respiratory, thoracic and mediastinal disorders) | 1 | 0
sinusitis (Infections and infestations) | 1 | 0
infection bladder (Infections and infestations) | 1 | 0
renal failure acute (Renal and urinary disorders) | 1 | 0
disease progression (General disorders) | 5 | 2
cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
thrombosis (Vascular disorders) | 0 | 2
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone 16 mg/m^2 (N=82) | Ixabepilone 40 mg/m^2 (N=89)
allergic reaction (Immune system disorders) | 5 | 6
neutropenia (Blood and lymphatic system disorders) | 15 | 47
anemia (Blood and lymphatic system disorders) | 12 | 31
thrombocytopenia (Blood and lymphatic system disorders) | 1 | 15
leucopenia (Blood and lymphatic system disorders) | 5 | 13
hypotension (Vascular disorders) | 2 | 6
weakness (General disorders) | 33 | 45
chills (General disorders) | 2 | 6
weight loss (Investigations) | 3 | 8
alopecia (Skin and subcutaneous tissue disorders) | 21 | 54
nail disorder (Skin and subcutaneous tissue disorders) | 9 | 5
rash (Skin and subcutaneous tissue disorders) | 9 | 9
constipation (Gastrointestinal disorders) | 20 | 20
dysguesia (Nervous system disorders) | 8 | 16
dehydration (Metabolism and nutrition disorders) | 4 | 14
vomiting (Gastrointestinal disorders) | 14 | 20
nausea (Gastrointestinal disorders) | 31 | 39
gastroesophageal reflux (Gastrointestinal disorders) | 2 | 8
diarrhea (Gastrointestinal disorders) | 18 | 19
mucositis (General disorders) | 3 | 10
abdominal pain (Gastrointestinal disorders) | 7 | 4
anorexia (Metabolism and nutrition disorders) | 17 | 24
infection fungal (Infections and infestations) | 1 | 6
fever (General disorders) | 8 | 13
edema (General disorders) | 11 | 12
hypokalemia (Metabolism and nutrition disorders) | 6 | 3
muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 13
pain bone (Musculoskeletal and connective tissue disorders) | 7 | 16
anxiety (Psychiatric disorders) | 3 | 6
neuropathy peripheral (Nervous system disorders) | 26 | 39
insomnia (Psychiatric disorders) | 8 | 9
headache (Nervous system disorders) | 13 | 13
dizziness (Nervous system disorders) | 10 | 15
neuropathy (Nervous system disorders) | 13 | 9 — For 13 participants in ixabepilone 16 mg/m2 group and 9 participants in ixabepilone 40 mg/m2 group, no detailed information indicated the 'neuropathy' as the 'peripheral neuropathy' or not.
pain (General disorders) | 23 | 27
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 13 | 15
pharyngitis (Infections and infestations) | 7 | 7
infection upper respiratory (Infections and infestations) | 4 | 9
cough (Respiratory, thoracic and mediastinal disorders) | 14 | 15
sinusitis (Infections and infestations) | 5 | 4
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5
infection bladder (Infections and infestations) | 5 | 7
myalgia (Musculoskeletal and connective tissue disorders) | 10 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.